CLINICAL TRIAL: NCT02525302
Title: HT-100 Long-term Safety and Pharmacodynamics in Patients With DMD Who Have Completed Protocols HALO-DMD-01 and HALO-DMD-02
Brief Title: HT-100 Long-term Study in DMD Patients Who Completed HALO-DMD-02
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Dosing stopped
Sponsor: Akashi Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HALO-DMD-03
Record Dates: First submitted 2015-07-18; First posted 2015-08-17 (Estimated); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: DMD; neuromuscular; Duchenne
MeSH Terms: conditions — Muscular Dystrophy, Duchenne | interventions — halofuginone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1: HT-100 tablet, Dose 1 (Experimental): HT-100 multiple dose administration (dose 1).
  Interventions: Drug: HT-100
- Cohort 1: HT-100 tablet, Dose 2 (Experimental): HT-100 multiple dose administration (dose 1).
  Interventions: Drug: HT-100
- Cohort 1: HT-100 tablet, Dose 3 (Experimental): HT-100 multiple dose administration (dose 1).
  Interventions: Drug: HT-100
- Cohort 1: HT-100 tablet, Dose 4 (Experimental): HT-100 multiple dose administration (dose 1).
  Interventions: Drug: HT-100
- Cohort 1: HT-100 tablet, Dose 5 (Experimental): HT-100 multiple dose administration (dose 1).
  Interventions: Drug: HT-100

INTERVENTIONS:
Drug: HT-100 — HT-100 is Akashi Therapeutics' proprietary delayed-release formulation of halofuginone hydrobromide, a small molecule therapeutic with anti-fibrotic properties. May be administered in either fed or fasted state. Not mutation specific.
  Other Names: halofuginone hydrobromide

SUMMARY:
This study, HALO-DMD-03, is a follow-on study to HALO-DMD-01 and HALO-DMD-02, and allows continued open-label access to HT-100 for subjects who have completed these studies. HALO-DMD-03 will provide safety and strength and function data on continuous long-term dosing. Data from this study will be used to inform the safety, tolerability, and dose selection for a future trial of HT-100 in boys with Duchenne Muscular Dystrophy (DMD).

DETAILED DESCRIPTION:
As a follow-on study to the initial clinical studies of HT-100 in DMD (Protocols HALO-DMD-01 and HALO-DMD-02), this open-label study is designed to provide data on continuous long-term dosing. Subjects will be entered into the study without cessation of dosing, in a staggered fashion, into the same cohort assignment they had in the predecessor studies. Up to 30 subjects who have completed dosing in HALO-DMD-02 will be offered the opportunity to continue on the same dose regimen until market approval of HT-100 or termination of the study by the Sponsor. Reasons for termination could include, among others, safety concerns or lack of efficacy, based on analysis of combined data from all HT-100 studies. Safety data from subjects approaching the end the HALO-DMD-02 participation will be individually reviewed by the Medical Monitor and the subject's physician (Principal Investigator [PI]). If the Medical Monitor and the PI agree there are no clinically significant safety signals (absence of clinically significant laboratory or clinical abnormalities to date), the subject will be considered eligible and offered continuation of dosing. To avoid an interruption in dosing, subjects will immediately be screened for participation and enrolled upon completing the predecessor trial, HALO-DMD-02. Participation is in this study HALO-DMD-03 is optional. Safety and pharmacodynamics (PD) monitoring will continue throughout the subject's study participation. Dose reduction/modification might occur or individual subjects' participation in the trial may be discontinued if any Adverse Events (AEs) suggest that HT-100 is not sufficiently well tolerated.

ELIGIBILITY:
Inclusion Criteria:

1. Completed both previous studies HALO-DMD-01 and HALO-DMD-02
2. Ability to provide written informed consent
3. Ability to understand and follow site and protocol instruction for the entire duration of the study

Exclusion Criteria:

Answering yes to any of the following make the subject NOT eligible to participate in the study.

1. Clinically significant major disease not related to DMD that would make it not safe to be in the study or affect ability to follow the protocol
2. History of severe allergic or anaphylactic reactions
3. Recent report of drug/alcohol abuse

Ages: 6 Years to 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2015-05; Primary Completion 2016-12-30 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Number of adverse events by severity and relationship | Every 6 months from enrollment for up to 3 years
Dose reduction or modification due to upper GI or other adverse events | Every 6 months from enrollment for up to 3 years
Trial discontinuations due to upper GI or other AEs | Every 6 months from enrollment for up to 3 years
Vital signs (Number of subjects with clinically significant changes) | Every 6 months from enrollment for up to 3 years
  Number of subjects with clinically significant changes
Laboratory values (Number of subjects with clinically significant changes) | Every 6 months from enrollment for up to 3 years
  Number of subjects with clinically significant changes.
Electrocardiograms | Every 6 months from enrollment for up to 3 years
  Number of subjects with clinically significant changes in QT interval
Echocardiograms | Every 6 months from enrollment for up to 3 years
  Number of subjects with clinically significant changes in left ventricular ejection fraction, end systolic and diastolic interventricular septal thickness, left ventricular posterior wall thickness
Cardiovascular Magnetic Resonance | Every 6 months from enrollment for up to 3 years
  Number of subjects with clinically significant change in diagnostic interpretation

SECONDARY OUTCOMES:
Cardiovascular Magnetic Resonance | Every 6 months from enrollment for up to 3 years
  Circumferential strain and myocardial fibrotic areas
Pulmonary function testing (Number of subjects with clinically significant changes) | Every 6 months from enrollment for up to 3 years
  Number of subjects with clinically significant changes.
Motor function measure (MFM) scale | Every 6 months from enrollment for up to 3 years
Performance of upper limb (PUL) scale | Every 6 months from enrollment for up to 3 years
Biomarkers of extracellular matrix turnover (Number of subjects with clinically significant changes) | Every 6 months from enrollment for up to 3 years
  Number of subjects with clinically significant changes.
Quantitative muscle testing (QMT) scores | Every 6 months from enrollment for up to 3 years
Timed function tests (TFTs) | Every 6 months from enrollment for up to 3 years
Motor Function Measure (MFM) | Every 6 months from enrollment for up to 3 years
Upper extremity function (proximal, mid-range, and distal) by Performance of Upper Limb (PUL) | Every 6 months from enrollment for up to 3 years
9-hole peg test | Every 6 months from enrollment for up to 3 years
  Assessment of upper limb function and dexterity
Tip pinch and key pinch tests (Number of subjects with clinically significant changes) | Every 6 months from enrollment for up to 3 years
  Number of subjects with clinically significant changes.
Electrical impedance myography (EIM) score | Every 6 months from enrollment for up to 3 years

OTHER OUTCOMES:
Pharmacokinetics peak plasma concentration (Cmax) | Pre-dose and 2-4 hour post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Diana M Escolar, MD, Study Director — Askashi Therapeutics
Locations (5):
- United States (5):
  - University of California, Davis Medical Center, Sacramento, California
  - Kennedy Krieger Institute, Johns Hopkins School of Medicine, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio

REFERENCES:
- See also: Sponsor company website — http://www.akashirx.com/